CLINICAL TRIAL: NCT01133600
Title: Phase IV Study of the Outpatient Treatment of Gram Positive Wound Infections in the Diabetic Foot: A Pharmaco-Economic Comparison of Daptomycin vs Vancomycin Based Regimens
Brief Title: Outpatient Treatment of Gram Positive Wound Infections in the Diabetic Foot: A Pharmaco-economic Comparison of Daptomycin vs. Vancomycin Based Regimens
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patient enrollment
Sponsor: Clinical Alliance for Research & Education - Infectious Diseases, LLC. (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Donald Poretz, Research Director, Clinical Alliance for Research & Education - Infectious Diseases, LLC.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0020-15
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- daptomycin (Active Comparator): Dosed at 6mg/kg body weight intravenously every 24 hours with a reduction to 6mg/kg every other day if creatinine clearance (CrCl)is <30ml/min.
  Interventions: Drug: Cubicin
- vancomycin (Active Comparator): Dosed at 15mg/kg intravenously every 12 hours with adjustments for renal function.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Cubicin — dosed at 6 mg/kg body weight intravenously every 24 hours with a reduction to 6mg/kg every other day if CrCl is <30ml/min.
  Arms: daptomycin
Drug: Vancomycin — dosed at 15mg/kg intravenously every 12 hours with adjustments for renal function.
  Arms: vancomycin

SUMMARY:
The purpose of the study is to evaluate the overall burden to the participant (economic, quality of life, patients satisfaction and freedom from side effects) when treating Gram positive infections of the foot in diabetic adults with daptomycin versus vancomycin.

DETAILED DESCRIPTION:
1. to compare the overall economic burden of therapy of a daptomycin vs. a vancomycin based antibiotic regimen for diabetic foot infections in the outpatient setting
2. to compare Quality of Life and patient satisfaction among recipients of a daptomycin vs. a vancomycin based regimen
3. to compare the safety and tolerance (adverse experiences) of daptomycin vs. vancomycin based regimens
4. to compare the efficacy (complete resolution of infection) of daptomycin vs. vancomycin based regimens

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 who are able to give informed consent and, who are likely to be able to participate through the full 28 day of the study.
* Previously diagnosed diabetes mellitus, requiring the use of insulin and/or oral hypoglycemic agents for glycemic control.
* The presence of an infection of one or both feet (defined as being distal to the superior-most point of the lateral malleolus), with some drainage, abscess or fluid collection that can be cultured, yet which as not been treated for greater than 24 hours with prior oral antibiotic therapy within the last 48 hours, wand which does not include either a quinolone or linezolid. The foot lesion, in the opinion of the initial treating physician, is severe enough (either because of the lesion or because of the subject's diabetic control, vasculopathy, etc) to require intravenous antibiotics.
* A culture of the wound, either at the time of screening or within the 72 hours prior to screening, that yields a Gram positive organism that is shown to be sensitive (or is likely to be sensitive) to both vancomycin and daptomycin. This will include Staphylococcus aureus, (including MSSA and MRSA, but excluding VRSA), Enterococcus faecalis and enterococcus faecium (excluding VRE), streptococci, including Groups A and B, as well as other beta-hemolytic streptococci, viridans streptococci, and Group D. A culture of coagulase negative staphylococci as the only Gram positive isolate will not be considered for participation. Cultures may be obtained as swab or fluid submitted for culture.
* Able to read and write in English with a proficiency suitable for completing the pharmaco-economic and quality of life questionnaires and diaries.

Exclusion Criteria:

* No Gram positive bacteria identified in the infected foot, infection with a Gram positive organism that is resistant to one of the two study drugs, or infection with coagulase negative staphylococci as the only Gram positive organism isolated.
* Known hypersensitivity to either of the two proposed study agents, or to ciprofloxacin, if a second anti-microbial agent is necessary.
* Renal dysfunction, such that the study subject requires dialysis.
* The presence of active osteomyelitis in the foot.
* The presence of concomitant infections that would require antibiotic therapy in addition to that being prescribed for the foot infection.
* The presence of pneumonitis requiring antimicrobial therapy, regardless of the suspected etiologic organism.
* A history of drug induced ototoxicity (either auditory or vestibular).
* A history of previous or current vascular catheter-associated phlebitis.
* Pregnancy or breastfeeding.
* Alcohol or drug use which, in the opinion of the investigator, is likely to interfere with the conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pharmaco-economic | 28 days
  Based upon 2 economic parameters associated with the treatment of the infection (provider charges and out-of-pocket costs) from screening until Day 28. Provider charges, as documented in invoices submitted to the pt's. insurance company, will be collected for all activities and services provided by the physician's office,home infusion company, laboratory, etc. during the study period. Out of pocket costs will be captured in a pt. diary and will include any health related costs that are borne by the pt. during the study period. Costs and charges will be analyzed and reported separately.

SECONDARY OUTCOMES:
Quality of Life/patient satisfaction | 28 days
  QOL and pt. satisfaction with the medication, the clinical care, and the overall experience of the infection and its therapy are captured using three study intstruments, which are described in more detail in the Data Collection Instruments section. These include two validated, standardized QOL instruments administred at Baseline, at two weeks and again at 4 weeks, and a pt. satisfaction survey administered at Baseline, 2 and 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Poretz, MD, Principal Investigator — Clinical Alliance for Research & Education - Infectious Diseases, LLC.
Locations (2):
- United States (2):
  - Clinical Alliance for Research & Education, Infectious Diseases, LlC, Annandale, Virginia
  - Infuscience, Annandale, Virginia